CLINICAL TRIAL: NCT00800111
Title: Open-enrollment, Prospective Study of Endothelial Keratoplasty Outcomes
Brief Title: Study of Endothelial Keratoplasty Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornea Research Foundation of America (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFA2008-01
Record Dates: First submitted 2008-11-26; First posted 2008-12-01 (Estimated); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Fuchs' Endothelial Corneal Dystrophy; Bullous Keratopathy; Iridocorneal Endothelial Syndrome; Posterior Polymorphous Dystrophy
Keywords: failed penetrating keratoplasty
MeSH Terms: conditions — Fuchs' Endothelial Dystrophy; Iridocorneal Endothelial Syndrome | interventions — Descemet Stripping Endothelial Keratoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Other): Endothelial keratoplasty procedure is performed.
  Interventions: Procedure: endothelial keratoplasty

INTERVENTIONS:
Procedure: endothelial keratoplasty — Endothelial keratoplasty is surgical replacement of the corneal endothelial cell layer (the cell layer lining the inner surface of the cornea).
  Other Names: Descemet stripping endothelial keratoplasty; Descemet stripping automated endothelial keratoplasty; Descemet membrane endothelial keratoplasty; DSEK; DSAEK; DMEK

SUMMARY:
Endothelial keratoplasty is a cornea-sparing transplant technique that replaces only the diseased endothelial cell layer of the patient's cornea. This technique offers many advantages compared with traditional full-thickness cornea transplants. Patients experience minimal change in glasses prescription and usually recover useful vision within weeks. Visual fluctuations are minimal during the healing process. The patient's cornea remains structurally intact and is more resistant to injury.

Endothelial keratoplasty is undergoing rapid and widespread adoption. Between 2005 and 2007, the number of corneas placed by US eye banks for endothelial keratoplasty increased ten-fold (2007 Eye Bank Association of America Annual Report). However, the procedure is less than 10 years old, and little is known about long term outcomes. Endothelial keratoplasty candidates at our center are invited to participate in an open enrollment, prospective study of the long-term outcomes of this procedure.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 or older
* Scheduled to undergo endothelial keratoplasty
* Able to provide written informed consent.

Exclusion Criteria:

* Age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2593 (Actual)
Dates: Start 2008-02; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 1, 3, 6, and 12 months and annually

SECONDARY OUTCOMES:
Endothelial cell density | 6 months, 12 months and annually
Intraocular pressure | 1, 3, 6, 12 months and annually
Manifest refraction | 1, 3, 6, 12 months and annually
corneal pachymetry | 1, 3, 6, 12 months and annually

CONTACTS AND LOCATIONS:
Overall Officials: Francis W Price, Jr., MD, Principal Investigator — Cornea Research Foundation of America
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Vajaranant TS, Price MO, Price FW, Wilensky JT, Edward DP. Intraocular pressure measurements following Descemet stripping endothelial keratoplasty. Am J Ophthalmol. 2008 May;145(5):780-6. doi: 10.1016/j.ajo.2008.01.010. Epub 2008 Mar 10. PMID 18329627
- [Background] Allan BD, Terry MA, Price FW Jr, Price MO, Griffin NB, Claesson M. Corneal transplant rejection rate and severity after endothelial keratoplasty. Cornea. 2007 Oct;26(9):1039-42. doi: 10.1097/ICO.0b013e31812f66e5. PMID 17893530
- [Background] Price MO, Price FW Jr. Endothelial cell loss after descemet stripping with endothelial keratoplasty influencing factors and 2-year trend. Ophthalmology. 2008 May;115(5):857-65. doi: 10.1016/j.ophtha.2007.06.033. Epub 2007 Sep 14. PMID 17868873
- [Background] Price MO, Price FW. Descemet's stripping endothelial keratoplasty. Curr Opin Ophthalmol. 2007 Jul;18(4):290-4. doi: 10.1097/ICU.0b013e3281a4775b. PMID 17568204
- [Background] Price MO, Price FW Jr, Trespalacios R. Endothelial keratoplasty technique for aniridic aphakic eyes. J Cataract Refract Surg. 2007 Mar;33(3):376-9. doi: 10.1016/j.jcrs.2006.10.052. PMID 17321384
- [Background] Price FW Jr, Price MO. Endothelial keratoplasty to restore clarity to a failed penetrating graft. Cornea. 2006 Sep;25(8):895-9. doi: 10.1097/01.ico.0000227888.03877.22. PMID 17102663
- [Background] Price MO, Price FW Jr. Descemet's stripping with endothelial keratoplasty: comparative outcomes with microkeratome-dissected and manually dissected donor tissue. Ophthalmology. 2006 Nov;113(11):1936-42. doi: 10.1016/j.ophtha.2006.05.034. Epub 2006 Aug 28. PMID 16935344
- [Background] Price FW Jr, Price MO. Descemet's stripping with endothelial keratoplasty in 200 eyes: Early challenges and techniques to enhance donor adherence. J Cataract Refract Surg. 2006 Mar;32(3):411-8. doi: 10.1016/j.jcrs.2005.12.078. PMID 16631048
- [Background] Price FW Jr, Price MO. Descemet's stripping with endothelial keratoplasty in 50 eyes: a refractive neutral corneal transplant. J Refract Surg. 2005 Jul-Aug;21(4):339-45. doi: 10.3928/1081-597X-20050701-07. PMID 16128330
- [Result] Guerra FP, Anshu A, Price MO, Giebel AW, Price FW. Descemet's membrane endothelial keratoplasty: prospective study of 1-year visual outcomes, graft survival, and endothelial cell loss. Ophthalmology. 2011 Dec;118(12):2368-73. doi: 10.1016/j.ophtha.2011.06.002. Epub 2011 Aug 27. PMID 21872938
- [Result] Pereira Cda R, Guerra FP, Price FW Jr, Price MO. Descemet's membrane automated endothelial keratoplasty (DMAEK): visual outcomes and visual quality. Br J Ophthalmol. 2011 Jul;95(7):951-4. doi: 10.1136/bjo.2010.191494. Epub 2010 Dec 22. PMID 21183511
- [Result] McCauley MB, Price MO, Fairchild KM, Price DA, Price FW Jr. Prospective study of visual outcomes and endothelial survival with Descemet membrane automated endothelial keratoplasty. Cornea. 2011 Mar;30(3):315-9. doi: 10.1097/ICO.0b013e3181eeb71b. PMID 21099412
- [Result] Guerra FP, Anshu A, Price MO, Price FW. Endothelial keratoplasty: fellow eyes comparison of Descemet stripping automated endothelial keratoplasty and Descemet membrane endothelial keratoplasty. Cornea. 2011 Dec;30(12):1382-6. doi: 10.1097/ICO.0b013e31821ddd25. PMID 21993468
- [Result] Kwon RO, Price MO, Price FW Jr, Ambrosio R Jr, Belin MW. Pentacam characterization of corneas with Fuchs dystrophy treated with Descemet membrane endothelial keratoplasty. J Refract Surg. 2010 Dec;26(12):972-9. doi: 10.3928/1081597X-20100212-08. Epub 2010 Feb 15. PMID 20166622
- [Result] Price MO, Giebel AW, Fairchild KM, Price FW Jr. Descemet's membrane endothelial keratoplasty: prospective multicenter study of visual and refractive outcomes and endothelial survival. Ophthalmology. 2009 Dec;116(12):2361-8. doi: 10.1016/j.ophtha.2009.07.010. Epub 2009 Oct 28. PMID 19875170
- [Result] McCauley MB, Price FW Jr, Price MO. Descemet membrane automated endothelial keratoplasty: hybrid technique combining DSAEK stability with DMEK visual results. J Cataract Refract Surg. 2009 Oct;35(10):1659-64. doi: 10.1016/j.jcrs.2009.05.034. PMID 19781456
- [Result] Feng MT, Burkhart ZN, Price FW Jr, Price MO. Effect of donor preparation-to-use times on Descemet membrane endothelial keratoplasty outcomes. Cornea. 2013 Aug;32(8):1080-2. doi: 10.1097/ICO.0b013e318292a7e5. PMID 23635858
- [Result] Anshu A, Price MO, Price FW Jr. Descemet stripping automated endothelial keratoplasty for Fuchs endothelial dystrophy-influence of graft diameter on endothelial cell loss. Cornea. 2013 Jan;32(1):5-8. doi: 10.1097/ICO.0b013e318247311a. PMID 22710494
- [Result] Anshu A, Price MO, Price FW Jr. Descemet membrane endothelial keratoplasty and hybrid techniques for managing failed penetrating grafts. Cornea. 2013 Jan;32(1):1-4. doi: 10.1097/ICO.0b013e3182488888. PMID 22710497
- [Result] Anshu A, Price MO, Price FW. Descemet's stripping endothelial keratoplasty: long-term graft survival and risk factors for failure in eyes with preexisting glaucoma. Ophthalmology. 2012 Oct;119(10):1982-7. doi: 10.1016/j.ophtha.2012.04.031. Epub 2012 Jun 15. PMID 22705345
- [Result] Anshu A, Price MO, Price FW Jr. Risk of corneal transplant rejection significantly reduced with Descemet's membrane endothelial keratoplasty. Ophthalmology. 2012 Mar;119(3):536-40. doi: 10.1016/j.ophtha.2011.09.019. Epub 2012 Jan 3. PMID 22218143
- [Result] Chaurasia S, Price MO, McKee Y, Price FW Jr. Descemet membrane endothelial keratoplasty combined with epithelial debridement and mitomycin-C application for fuchs dystrophy with preoperative subepithelial fibrosis or anterior basement membrane dystrophy. Cornea. 2014 Apr;33(4):335-9. doi: 10.1097/ICO.0000000000000078. PMID 24488132
- [Result] Chaurasia S, Price FW Jr, Gunderson L, Price MO. Descemet's membrane endothelial keratoplasty: clinical results of single versus triple procedures (combined with cataract surgery). Ophthalmology. 2014 Feb;121(2):454-8. doi: 10.1016/j.ophtha.2013.09.032. Epub 2013 Nov 16. PMID 24252821
- [Result] Feng MT, Price MO, Miller JM, Price FW Jr. Air reinjection and endothelial cell density in Descemet membrane endothelial keratoplasty: five-year follow-up. J Cataract Refract Surg. 2014 Jul;40(7):1116-21. doi: 10.1016/j.jcrs.2014.04.023. PMID 24957432
- [Result] Burkhart ZN, Feng MT, Price FW Jr, Price MO. One-year outcomes in eyes remaining phakic after Descemet membrane endothelial keratoplasty. J Cataract Refract Surg. 2014 Mar;40(3):430-4. doi: 10.1016/j.jcrs.2013.08.047. Epub 2014 Jan 11. PMID 24417895
- [Result] Schoenberg ED, Price FW Jr, Miller J, McKee Y, Price MO. Refractive outcomes of Descemet membrane endothelial keratoplasty triple procedures (combined with cataract surgery). J Cataract Refract Surg. 2015 Jun;41(6):1182-9. doi: 10.1016/j.jcrs.2014.09.042. Epub 2015 Jun 19. PMID 26096520
- [Result] Price MO, Feng MT, McKee Y, Price FW Jr. Repeat Descemet Membrane Endothelial Keratoplasty: Secondary Grafts with Early Intervention Are Comparable with Fellow-Eye Primary Grafts. Ophthalmology. 2015 Aug;122(8):1639-44. doi: 10.1016/j.ophtha.2015.04.037. Epub 2015 Jun 6. PMID 26050537
- [Result] Tenkman LR, Price FW, Price MO. Descemet membrane endothelial keratoplasty donor preparation: navigating challenges and improving efficiency. Cornea. 2014 Mar;33(3):319-25. doi: 10.1097/ICO.0000000000000045. PMID 24452215
- [Result] Price MO, Lisek M, Feng MT, Price FW Jr. Effect of Donor and Recipient Diabetes Status on Descemet Membrane Endothelial Keratoplasty Adherence and Survival. Cornea. 2017 Oct;36(10):1184-1188. doi: 10.1097/ICO.0000000000001305. PMID 28749899
- [Result] Gonzalez A, Price FW Jr, Price MO, Feng MT. Prevention and Management of Pupil Block After Descemet Membrane Endothelial Keratoplasty. Cornea. 2016 Nov;35(11):1391-1395. doi: 10.1097/ICO.0000000000001015. PMID 27560030
- [Result] Price DA, Price MO, Lopez A, Price FW Jr. Effect of Descemet Membrane Endothelial Keratoplasty on Color Vision in Patients With Fuchs Dystrophy. Cornea. 2016 Aug;35(8):1045-8. doi: 10.1097/ICO.0000000000000871. PMID 27158810
- [Result] Price MO, Calhoun P, Kollman C, Price FW Jr, Lass JH. Descemet Stripping Endothelial Keratoplasty: Ten-Year Endothelial Cell Loss Compared with Penetrating Keratoplasty. Ophthalmology. 2016 Jul;123(7):1421-7. doi: 10.1016/j.ophtha.2016.03.011. Epub 2016 Apr 20. PMID 27108095
- [Result] Price MO, Scanameo A, Feng MT, Price FW Jr. Descemet's Membrane Endothelial Keratoplasty: Risk of Immunologic Rejection Episodes after Discontinuing Topical Corticosteroids. Ophthalmology. 2016 Jun;123(6):1232-6. doi: 10.1016/j.ophtha.2016.02.001. Epub 2016 Mar 13. PMID 26983976
- [Result] Crews JW, Price MO, Lautert J, Feng MT, Price FW Jr. Intraoperative hyphema in Descemet membrane endothelial keratoplasty alone or combined with phacoemulsification. J Cataract Refract Surg. 2018 Feb;44(2):198-201. doi: 10.1016/j.jcrs.2017.11.015. Epub 2018 Mar 7. PMID 29525615
- [Result] Price DA, Kelley M, Price FW Jr, Price MO. Five-Year Graft Survival of Descemet Membrane Endothelial Keratoplasty (EK) versus Descemet Stripping EK and the Effect of Donor Sex Matching. Ophthalmology. 2018 Oct;125(10):1508-1514. doi: 10.1016/j.ophtha.2018.03.050. Epub 2018 May 3. PMID 29731147
- See also: Cornea Research Foundation of America website — http://www.cornea.org